CLINICAL TRIAL: NCT04781660
Title: A Clinical Research for Safety and Feasibility of Implantable Alginate Hydrogel as a Method of Left Ventricular Restoration in Patients With Heart Failure
Brief Title: First in Man Study of Implantable Alginate Hydrogel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK/CQ/CM-001-CIP-01
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: caused by ischemic cardiomyopathy; caused by non-ischemic cardiomyopathy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantable Alginate Hydrogel (Experimental): All patients will be treated with Implantable Alginate Hydrogel
  Interventions: Device: Implantable Alginate Hydrogel

INTERVENTIONS:
Device: Implantable Alginate Hydrogel — Implantable Alginate Hydrogel is a single use, multiple component device. It is expected to be used as a space-occupying material implanted into the myocardium to affect the shape of the left ventricle and reduce the clinical symptoms of patients with left ventricular ischemia and non-ischemic cardiomyopathy.
  The hydrogel serves as an artificial myocardial filler to stop the continuous expansion of the ventricle and restore it to a more favorable shape and size. The expected clinical effect of the Implanted Alginate Hydrogel is to reduce the clinical symptoms of patients and improve the quality of life by improving the structure and function of the failing heart.

SUMMARY:
The objective of this clinical research is to evaluate the safety and effectiveness of Implantable Alginate Hydrogel to reconstruct the left ventricle in the treatment of heart failure

ELIGIBILITY:
Inclusion Criteria:

1. The patients must have been able and willing to give written informed consent
2. The patients should be adult (age≥ 18 years and <75 years) males or females
3. The patients must have been on stable, evidence-based therapy for HF
4. The Patients have a LVEF ≤35%
5. NYHA is classified as grade III or IV
6. If female, the patients must have been (a) post-menopausal, (b) surgically sterile, or (c) using adequate birth control and have a negative serum pregnancy test within 7 days prior to administration of the study device.

Exclusion Criteria:

1. Have undergone any therapeutic traumatic heart surgery within 30 days.
2. Hemodynamic instability or cardiogenic shock.
3. Right-sided HF.
4. Patients who presented with a restrictive cardiomyopathy such as due to amyloidosis, sarcoidosis, or hemochromatosis.
5. History of Constrictive pericarditis.
6. History of stroke (within 60 days prior to the surgical procedure).
7. History of myocardial infarction (within 30 days prior to the surgical procedure).
8. An LV wall thickness of the LV free-wall, at the mid-ventricular level, of < 6 mm.
9. Serum creatinine > 2.0 mg/dL, or calculate creatinine clearance rate <25 mL/min
10. Clinically significant liver enzyme abnormalities, i.e., aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 2 times the upper limit of normal and/or bilirubin more than 50% above the upper limit of normal.
11. Had been receiving concurrently an investigational product in another clinical trial or had received an investigational product in another clinical trial in the 30 days prior to enrollment.
12. A life expectancy of < 1 year due to comorbidities .
13. Unfit for the minimal invasive treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Device Events | 30 days after implantation
  Definition of SADE: Any complications related to the device include but not limited: death, stroke, permanent damage to the heart, any situation that requires further intervention, etc.

SECONDARY OUTCOMES:
Device successfully Setup rate | immediately after the implantation
  Device successfully Setup defined as:
  1. The device reaches the expected implant location
  2. Implant the hydrogel accurately in the left ventricle wall for 6~12 implant points.
  3. Remove the delivery system
Incidence of SAE | Within 6 months after implantation
  Rate of Serious Adverse Events occurred during procedure and follow-up
NHYA Class level changes rate between baseline and 6 months' follow-up | 6 months after implantation
Quality of life changes rate between baseline and 6 months' follow-up | 6 months after implantation
Rate of Rehospitalization due to heart failure | within 6 months after implantation
  Rehospitalization due to heart failure within 6 months after implantation
LVEF changes rate between baseline and 6 months' follow-up | 6 months after implantation
Size of LV changes rate between baseline and 6 months' follow-up | 6 months after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Professor, Principal Investigator — The First Affiliated Hospital of Air Force Military Medical University
Locations (1):
- The First Affiliated Hospital of Air Force Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No